CLINICAL TRIAL: NCT07062016
Title: MC230601 Molecular and ctDNA Characterization of High-Risk Endometrial Cancer
Brief Title: Molecular and ctDNA Characterization of High-Risk Endometrial Cancer
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 25-000815; NCI-2025-04532 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 25-000815 (Other: Mayo Clinic Institutional Review Board); MC230601 (Other: Mayo Clinic)
Record Dates: First submitted 2025-07-02; First posted 2025-07-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Endometrial Carcinoma; Endometrial High Grade Endometrioid Adenocarcinoma; Stage II Endometrial Cancer; Stage III Endometrial Cancer; Stage IV Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Patients undergo blood and tissue sample collection and have their medical records reviewed throughout the study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study seeks to better understand the recurrence of high-risk endometrial cancer. It will collect information about cancer genetics to find out various hereditary or cancer specific genetic variants that may have a role in diagnosis or management and prognosis of cancer. It also seeks to develop a genetic results and medical record databank for future studies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To generate preliminary data for a risk stratification model for recurrence including traditional histopathologic risk factors, molecular characterization in endometrial cancer patients with features of aggressive disease.

OUTLINE: This is an observational study.

Patients undergo blood and tissue sample collection and have their medical records reviewed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Planned complete surgical staging at Mayo Clinic. Complete surgical staging includes at least total hysterectomy, bilateral salpingo-oophorectomy and lymph node assessment. Sentinel node mapping meets the criteria for lymph node assessment. Peritoneal cytology is recommended. Additional staging procedures such as pelvic and para-aortic nodal evaluation, omental biopsy or omentectomy, may also be utilized for staging in patients based on the clinical situation and at the surgeon's discretion
* At least one preoperative or postoperative feature of aggressive disease [International Federation of Gynecology and Obstetrics (FIGO) staging used throughout this protocol]

  * Preoperatively:

    * Biopsy with grade 3 endometrioid endometrial cancer (EC) or non-endometrioid EC
    * Patients with FIGO grade 1-2 EC with evidence of extrauterine disease on imaging (CT, MRI, or PET)
  * Postoperatively:

    * Endometrial cancer (FIGO) with one or more established risk factors:

      * Non-endometrioid histology

        * Grade 3
      * Lymphovascular space invasion (LVSI), ≥ 50% of myometrial invasion, presence of isolated tumor cells (ITC) in a sentinel lymph node OR
      * Stage II to IV (FIGO) EC
* Provide written informed consent
* Willingness to provide mandatory blood specimens for correlative research
* Willingness to provide mandatory tissue specimens for correlative research
* Willingness to return to registering site for clinical follow-up

Exclusion Criteria:

* Patient receiving or who has received neoadjuvant chemotherapy
* Pre-operative pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Endometrial cancer patients with aggressive disease and planned complete surgical staging at Mayo Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival (RFS) | Up to 3 years
  Defined as time from primary staging surgery to recurrence or death.
Presence of somatic and germline pathogenic variants | Up to 3 years
  For each participant, a surgical tissue sample (OncoExtra) and a presurgical blood sample (RiskGuard) sample will be utilized to determine the presence of somatic and germline pathogenic variants. The count and percentage of patients with the presence of somatic or germline variants will be reported by The Cancer Genome Atlas (TGCA) class. The number, type, and function of somatic variants will also be reported by TGCA class. For genes with alterations seen in at least 10 patients, a log rank test will be used to assess whether RFS differs with respect to whether an alternation is present or not.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Mariani, MD, MS, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials